CLINICAL TRIAL: NCT01965808
Title: Effect of Food on the Pharmacokinetics of LY2157299 Monohydrate in Healthy Subjects
Brief Title: A Study of LY2157299 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15239; H9H-MC-JBAU (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — LY-2157299

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2157299 (Fasted) (Experimental): Single dose of 150 mg LY2157299 administered orally in fasted state in one of two study periods.
  Interventions: Drug: LY2157299
- LY2157299 (Fed) (Experimental): Single dose of 150 mg LY2157299 administered orally in fed state in one of two study periods.
  Interventions: Drug: LY2157299

INTERVENTIONS:
Drug: LY2157299 — Administered orally

SUMMARY:
Participants in this study will receive two oral doses of 150 milligram (mg) LY2157299 taken at least 4 days apart. One dose will be given without food. One dose will be given with a high fat meal. The study will evaluate the effect of a high fat meal on how much of the drug gets into the blood stream. Side effects will be documented. This study will last approximately 15 days not including screening. Screening is required within 30 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy sterile males or females
* Are able to eat a high fat meal
* No abnormal heart function or high blood pressure
* No participation in a clinical trial within 30 days
* No evidence of human deficiency virus (HIV), hepatitis C or hepatitis B

Exclusion Criteria:

* Have a clinically significant abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum Concentration (Cmax) of LY2157299 | Pre-dose through 72 hours post-dose in each study period
Pharmacokinetics: Time of Maximum Observed Concentration (tmax) of LY2157299 | Pre-dose through 72 hours post-dose in each study period
Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY2157299 | Pre-dose through 72 hours post-dose in each study period

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States